CLINICAL TRIAL: NCT03678519
Title: Occupational Health Hazards Among Flour Mills Workers And Smoking Situation Analysis Among Smokers, Assiut
Brief Title: Occupational Health Hazards Among Flour Mills Workers
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ayah Atef Alkarn, Principal investigator, Assiut University
Other Study IDs: OHHFM
Record Dates: First submitted 2018-09-17; First posted 2018-09-19 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Occupational Exposure
MeSH Terms: interventions — Respiratory Function Tests

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Exposed workers: Flour mills workers exposed to health hazards
  Interventions: Diagnostic Test: Pulmonary function test

INTERVENTIONS:
Diagnostic Test: Pulmonary function test — Pulmonary Function tests using Spirometry. It will show following indices of ventilatory functions: Forced vital capacity (FVC), Forced expiratory volume in the 1st second (FEV1) and Forced expiratory volume in the 1st second as a percentage of the Forced vital capacity (FEV1/FVC %).

SUMMARY:
Flour milling is from the oldest trade industry. Several problems arise during functioning and maintenance operations. Production process involves the breakdown of grains to separate their outer covering and inner endosperm grinding to fine flour particles. Workers are at substantial risk with two main problems causing severe health issues and accidents. The first is the improper flour milling process including intake and final products collection systems. The second is the unawareness and unavailability of PPE.

DETAILED DESCRIPTION:
Flour is a complex organic dust consisting of one or a mixture of several cereal grains (wheat, rye, millet, barley, oats or corn cereal) that have been processed or ground by milling. In addition, flour may contain a diverse number of contaminants, such as silica, fungi and their metabolites (mycotoxins), bacterial endotoxins, insects, mites, mammalian debris and chemical additives such as pesticides and herbicides. Occupational exposure to flour dust occurs in different settings, as: bakeries, grain mills and flour mills.

Many industries, including flour mills, generate dust, which is released into air, then inhaled during industrial processes as: cleaning, packaging and shipping. Occupational respiratory diseases are usually caused by extended exposure to irritating or toxic substances that may cause acute or chronic respiratory diseases.

It has long been known that occupational exposure to flour dust may cause respiratory illness, ranging from simple irritation to rhinitis and asthma, due to components of the grains themselves as well as contaminants of the flour dust and additives.

Flour mills workers have been in an environment exposed to flour dust, suffering from sensitization, occupational asthma, allergic rhinitis, obstructive lung diseases and eye infection.

Mill workers' suffer from conjunctivitis, allergic and baker's asthma, wheezing, febrile reactions, grain fever, lung fibrosis, rhinitis, allergic alveolitis, impairment of lung function and chronic obstructive pulmonary disease. These respiratory symptoms with continuing occupational exposure can lead to worker disability that force them to leave their jobs.

Respiratory system symptoms and diseases induced by occupational dust are influenced by the type of dust, dose, duration of exposure and genetic factors.

A study carried out in Sohag found that respiratory symptoms were significantly higher among exposed workers as compared to unexposed. Furthermore a highly significant decline in pulmonary function tests.

The albumin portion of flour is the main cause of allergies that known as "Baker's asthma" (BA) and inhaling it leads to the stimulation of the specific antibodies, increased allergies, respiratory disorders and ultimately asthma.

Baker's asthma is one of the first occupational diseases described in the literature. Baker's asthma and baker's rhinitis are mainly due to type I sensitization to wheat. Studies demonstrate dose-response relationships between the exposure to wheat and the prevalence of immediate-type I sensitization or lung function impairments.

It was found that host and environmental factors play a role in asthma development. Environmental factors include: allergens either indoor or outdoor, infections, tobacco smoke, air pollution and occupational sensitizers.

Asthma caused by flour dust is described with a latent period between first exposure and development of symptoms, which varies from a few weeks to 35 years.

A relationship is present between asthma symptoms and the workplace in the form of: appearance of asthma symptoms at work or early night after returning home. It worsens at early night before sleep and improve or disappear at late night or early morning. Occupational asthma (OA) shows diurnal improvement of symptoms in contradictory to ordinary bronchial asthma. Also there is improvement of asthma away from work in the weekend and holidays and worsening of symptoms on returning to work showing weekly variability.

A study carried out in Helwan, showed that 25% of mills workers had asthma related to work. The asthma symptoms appear during work which showed improvement after leaving workplace. It showed also reversibility in FEV and diurnal PEFR variability. Also asthmatic workers had lower level of spirometric parameters.

Smoking, as an occupational hazard, has been studied extensively since the 1970s. For many, smoking is perceived as a coping strategy to mitigate work-related stress.

The tobacco epidemic is one of the biggest public health threats the world has ever faced. Smoking is the single largest cause of preventable death and disease killing more than 7 million people a year. More than 6 million of those deaths are the result of direct tobacco use while around 890 000 are the result of non-smokers being exposed to second-hand smoke. It is expected to increase to more than 8 million a year by 2030. Around 100 million people died because of tobacco use in the 20th century, and it will kill 1 billion people in the 21st century if current trends continue.

Smoking increases the risk for all-cause mortality and has been found to increase risk for various types of cancer, respiratory, cardiovascular, eye diseases, diabetes, impaired immune function and erectile dysfunction in men. Smoking may be a risk factor for high frequency hearing loss, and its combined effect on hearing with exposure to occupational noise is additive.

There are more than 4000 chemicals in tobacco smoke, of which at least 250 are known to be harmful and more than 50 are known to cause cancer.

Egypt is one of 15 countries worldwide with heavy burden of tobacco-related ill health. Egypt is also considered the leading Arab country in terms of tobacco-related deaths. About 40.5% of men are daily tobacco smokers. And, 49.9% of men according to Tobacco Atlas.

There is disparity in tobacco use between people of lower and higher socioeconomic status. Around 80% of the smokers live in low- and middle-income countries. People with less education and living in poor neighborhoods are associated with high risk of smoking.

A major concern is the Second-hand smoke (SHS) exposure, also known as ''involuntary smoking'' or ''passive smoking'', refers to non-smokers' inhalation of smoke from the exhalation of smokers or burning cigarettes. SHS contains hundreds of toxic and carcinogenic substances and related to many diseases as those of smokers. In Egypt, among those who worked indoors or in enclosed areas, 60.7% were exposed to second-hand smoke at work, including 58.5% non-smokers.

Smoking is Costing the workplace as a result of employee smoking. It costs employers more to employ smokers. These costs are primarily attributed to:

* Decreased productivity
* Increased absenteeism
* Workdays lost due to illnesses provoked or aggravated by smoking
* Unproductive time, such as smoke breaks
* Higher insurance premiums. Smoking cessation greatly diminishes the high risk of death. Stopping smoking improve life expectancy, reduce morbidity and costs associated with treating smoking related conditions. Smokers have shorter life than non-smokers. However, cessation will gradually reverse health risks associated with smoking, especially in younger individuals.

An assessment should reveal the level of motivation or 'stage of change' the employees at for smoking cessation. Employees may be in one of five stages of the stop smoking process. Pre-Contemplation, Contemplation, Preparation, Action and Maintenance. Smoking cessation could be conceptualized into two stage; first making a quit attempt, then succeeding in maintaining it.

Most adults spend approximately one-third of their day in a workplace, it can be a useful setting through which large groups of employees can be reached. Workplace smoking cessation interventions have positive effects and should be encouraged and promoted by health and work authorities. They help to increase the number of ex-smokers, those who continue smoking smoke fewer cigarettes and for nonsmoking workers, the workplace might be the only contact with tobacco smoke.

Quit rates in intervention groups are higher than in control groups in number of studies. Quit rates in intervention between 6.1-30.8% vs. 1.0-19.1% in control groups.

The workplace as a setting for smoking cessation research and intervention has several advantages:

1. It provides access to a large number of people which constitute a relatively stable population.
2. It has the potential for reaching a larger proportion of the smoking population than non-workplace environments.
3. Worksites have potential to provide sustained peer group support and positive peer influence for quitting and staying tobacco free.
4. It provides a particular opportunity to target young men, who traditionally have low general practitioner consultation rates and are thus less likely to benefit from health promotion activity.
5. Occupational health staff may be on hand to give professional support.
6. The convenience of cessation programs onsite has an advantage to the employee.
7. Employers benefit from supporting employees for smoking cessation including increased productivity.

Having smoking friends and associates tends to make quitting more difficult, while smokers whose friends, coworkers, and family are former smokers are more likely to succeed in their attempts to quit smoking. Long term success was significantly better if more work-mates from the same department participated in the smoking cessation program.

Quitting behaviors were influenced by occupational class. Workers in blue-collar occupations such as in construction and maintenance are significantly more likely to be smokers than workers in white-collar occupations; those who work in office administration or in financial operations. White-collar workers are more likely to be influenced positively by anti-smoking programs than blue collars.

The task of the occupational physician is to inform workers about the high risks linked to smoking, passive smoking and obligations enforced by law, collect information about workers' smoking habits and promote smoking cessation.

ELIGIBILITY:
Workers in flour mills

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Flour Mills Workers, Assiut
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Detect number of workers who have occupational diseases | 6 months

SECONDARY OUTCOMES:
Number of patients who have declined pulmonary function tests | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nieva G, Comin M, Valero S, Bruguera E. Cigarette dependence and depressive symptoms as predictors of smoking status at five-year follow-up after a workplace smoking cessation program. Addict Behav. 2017 Oct;73:9-15. doi: 10.1016/j.addbeh.2017.04.003. Epub 2017 Apr 3. PMID 28431293
- [Background] Meo SA, Al-Drees AM. Lung function among non-smoking wheat flour mill workers. Int J Occup Med Environ Health. 2005;18(3):259-64. PMID 16411565
- [Background] Neghab M, Soltanzadeh A, Alipour A, Hasanzadeh J, Alipour H. Respiratory morbidity induced by occupational inhalation exposure to high concentrations of wheat flour dust. Int J Occup Saf Ergon. 2012;18(4):563-9. doi: 10.1080/10803548.2012.11076960. PMID 23294661
- [Background] Wang CP, Ma SJ, Xu XF, Wang JF, Mei CZ, Yang GH. The prevalence of household second-hand smoke exposure and its correlated factors in six counties of China. Tob Control. 2009 Apr;18(2):121-6. doi: 10.1136/tc.2008.024836. Epub 2009 Jan 8. PMID 19131456
- [Background] Fouad H, Awa FE, Naga RA, Emam AH, Labib S, Palipudi KM, Andes LJ, Asma S, Talley B. Prevalence of tobacco use among adults in Egypt, 2009. Glob Health Promot. 2016 Jun;23(2 Suppl):38-47. doi: 10.1177/1757975913499801. Epub 2013 Sep 16. PMID 24042971
- [Background] Abdullah AS, Driezen P, Quah AC, Nargis N, Fong GT. Predictors of smoking cessation behavior among Bangladeshi adults: findings from ITC Bangladesh survey. Tob Induc Dis. 2015 Aug 11;13(1):23. doi: 10.1186/s12971-015-0050-y. eCollection 2015. PMID 26261450
- [Background] Brown CRH, Forster S, Duka T. Goal-driven attentional capture by appetitive and aversive smoking-related cues in nicotine-dependent smokers. Drug Alcohol Depend. 2018 Sep 1;190:209-215. doi: 10.1016/j.drugalcdep.2018.06.011. Epub 2018 Jul 19. PMID 30055425
- [Background] Massin N, Bohadana AB, Wild P, Kolopp-Sarda MN, Toamain JP. Airway responsiveness to methacholine, respiratory symptoms, and dust exposure levels in grain and flour mill workers in eastern France. Am J Ind Med. 1995 Jun;27(6):859-69. doi: 10.1002/ajim.4700270609. PMID 7645579